CLINICAL TRIAL: NCT01014897
Title: tDCS in Chronic Stroke Recovery-pilot
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Chronic Stroke Recovery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 032009-067; 092010-231 (Other: UTSW IRB)
Record Dates: First submitted 2009-11-02; First posted 2009-11-17 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Stroke
Keywords: stroke; recovery; tDCS; direct current; electric stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- subcortical (Experimental): Subcortical stroke patients will receive tDCS stimulation and sham in random order
  Interventions: Device: tDCS
- cortical (Experimental): subjects will receive active and sham tDCS in random order
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS and sham will be applied in random order during standardized occupational therapy
  Other Names: transcranial direct current stimulation

SUMMARY:
The hypothesis of this study is that different subgroups of stroke will respond differently to direct current stimulation.

DETAILED DESCRIPTION:
We have tested the effectiveness of each stimulation condition: 1) anodal over the lesional motor cortex 2) anodal PMD (positive electrode at the dorsal premotor cortex (PMD) of the lesional hemisphere (first phase) or dual motor cortex stimulation (second phase), 3) cathodal over the contralesional motor cortex, and 4) sham in a double blind crossover design in chronic cortical and subcortical strokes.

Persons in the chronic stage of recovery from stroke (>3 months) will receive each type of tDCS stimulation for 20 minutes concurrent with physical therapy treatments (90 minutes ) utilizing the Armeo ®, a gravity neutral arm exercise support system for the most involved upper extremity which provides for task practice in a virtual reality environment, followed by a therapist supervised targeted hand exercise. The experimental protocol will not alter standard of care, will be performed after standard rehabilitation is completed. The experimental therapy is not part of standard care and will not be charged or reimbursed by the patients' insurance. Participation will be free of charge for subjects.

We were planning to perform the study in two phases. In the first exploratory phase, we will conduct a short pilot study with 15 subjects to optimize and if possible simplify the treatment parameters for the second longer phase of the experiment. In this first phase we will perform one of the four different tDCS stimulation conditions concurrently with the physical therapy protocol on each therapy day, so that all subjects will receive all stimulation types in a randomized counterbalanced order. There will be a 1 day rest period in between sessions, making 9 days (10 days if initial evaluation is done on the day before the 1st treatment) the total commitment time for the first phase of study.

The outcome measures were collected before and after each session. The outcome measures collected after the 1 day rest provide the baseline for the next session will be also used as to validate the stability of the treatment effect. Subjects participating in the first part of the study will be offered the option to participate in the second longer phase of the study. (please see table under study procedures)

In the second phase of the experiment we will perform only the promising stimulation paradigms plus sham from the first part of the experiment in a random, counterbalanced order on up to 30 chronic stroke subjects. If in the initial phase there are no differences found between stimulation types in the cortical vs subcortical patient groups then all 3 stimulation paradigms will be performed in the second phase.

Based on our preliminary data, we will perform the following paradigms in the second phase: 1) sham 2) dual stimulation 3) optimized tDCS in a randomized counterbalanced order. The optimized tDCS will be determined during a test session prior to the first treatment where the tDCS montage producing the best behavioral response will be used during therapy. Subjects will perform this under IRB approved study # STU 102013-085.

The patient time commitment in the second phase is 18 weeks, where subjects will have 3 x 1 weeks long treatment (5 weekdays) sessions with 5 week inter-treatment "rest period". The blinded tester will perform a final outcome evaluation 5 weeks after the end of the last session. (please see table under study procedures)

Total number of potential enrolled subjects for both phases will be approximately 45 [Phase 1 (15) + Phase 2 (30)].

The stepwise design will enable us to optimize study time commitment and expenses for both patients and researchers while maximizing clinical/scientific gain.

ELIGIBILITY:
Inclusion Criteria:

* single symptomatic stroke more than 3 months ago with hand/arm weakness
* able to perform required tests and provide consent
* Age 18-80
* Modified Ashworth scale <3
* range of motion functional at shoulder elbow wrist and hand

Exclusion Criteria:

* more than one symptomatic stroke in middle cerebral artery territory or bilateral involvement
* severe medical or psychiatric conditions, drug abuse, seizure disorder
* pregnancy/breast feeding
* subarachnoid hemorrhage, lobar hemorrhage
* patients who can not have tDCS (prior head surgery, pacemakers, metallic implants in the head etc)
* patients taking antiadrenergic medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function test | immediately before and immediately after treatment
  The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks. The WMFT has been posited as instructive for assessing the motor status of higher functioning chronic patients with stroke and traumatic brain injury, in terms of severity and upper extremity motor deficiency. The final time score will be the median time required for all timed tasks executed. One hundred twenty seconds is the maximum time allowed for each task attempted. Since medians will be used, all scores above the median (whether, e.g., 62 sec. or 120+ sec.) have the same weight
Fugl-Meyer Assessment | immediately before and immediately after treatment
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226, though it is common practice to assess all domains separately <50 = severe impairment, 50-84 = marked impairment, 85-94 = moderate impairment, 95-99= slight impairment

CONTACTS AND LOCATIONS:
Overall Officials: Timea Hodics, M.D., Principal Investigator — UTSW
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Derived] Hodics TM, Nakatsuka K, Upreti B, Alex A, Smith PS, Pezzullo JC. Wolf Motor Function Test for characterizing moderate to severe hemiparesis in stroke patients. Arch Phys Med Rehabil. 2012 Nov;93(11):1963-7. doi: 10.1016/j.apmr.2012.05.002. Epub 2012 May 10. PMID 22579647